CLINICAL TRIAL: NCT05409456
Title: Comparative Effects of Mild and Moderate Aerobic Exercises on Blood Pressure, Oxygen Saturation and Heart Rate in Hypertensive Patients
Brief Title: Comparative Effects of Mild and Moderate Aerobic Exercises on BP, VO2 and HR in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC/22/0330 Marryam
Record Dates: First submitted 2022-05-26; First posted 2022-06-08 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Hypertension
Keywords: HTN hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: two groups group A is assign mild aerobic group b is assign moderate aerobic
Who Masked: Outcomes Assessor
Masking Description: assessor is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mild aerobic exercise (Experimental): group A was given mild aerobic exercise on treadmill with warm up exercise
  Interventions: Other: mild aerobic exercise
- moderate aerobic exercise (Experimental): group B was moderate aerobic on treadmill with warm up exercise
  Interventions: Other: moderate aerobic exercise

INTERVENTIONS:
Other: mild aerobic exercise — mild aerobic exercise given to group A on treadmill
  Other Names: aerobic
  Arms: mild aerobic exercise
Other: moderate aerobic exercise — moderate aerobic exercise given to group B on treadmill
  Other Names: aerobic
  Arms: moderate aerobic exercise

SUMMARY:
World Health Organization, when systolic blood pressure is equal to or above 130 mm Hg and/or a diastolic blood pressure equal to or above 85 mm Hg , the blood pressure is considered to be raised or high is called hypertension." Most people with hypertension have no symptoms at all; this is why it is known as the "silent killer".

More than 1 in 5 adults worldwide had raised blood pressure. There has been studies on strength exercise, severe aerobic exercise and other types of exercises and on their effects on blood pressure, heart rate and oxygen saturation in other patient populations and on healthy individuals as well, but in the patients with hypertension no comparison has been made between mild and moderate aerobic exercise (tread mill) yet, stating which one is effective. Secondly, already present studies have shown long term effects mostly, not the comparative effects of mild and moderate exercises on blood pressure heart rate and oxygen saturation of patients with hypertension. These techniques are inexpensive, easy to perform and contain no known harmful effect. Hence, current study will undertake this task of finding out what are the comparative effects of mild and moderate aerobic on the BP, heart rate and oxygen saturation and secondly which technique is more effective. Study design will Randomized clinical trial with non-probability convenient sampling.

It will be single blinded study with blinding of assessor. Sample size was calculated from Epitools website and will be 28. There will be two groups which will be randomly assigned 14 people using lottery method. Data will be collected from community dwelling areas of Lahore Patients with hypertension with Systolic Blood Pressure 130 - 159 mmHg and Diastolic Blood Pressure 85 - 99 mmHg (pre hypertensive and stage 1), 30 to 50 years of age, patients who have taken any antihypertensive medicine in more than 6 hours and both males and females will be recruited. Tools will be aneroid sphygmomanometer for measuring blood pressure and pulse oximeter for measuring oxygen saturation and heart rate and Post interventional BP, heart rate readings and oxygen saturation will be taken for both groups on the same day.

Post intervention blood pressure, Heart rate and oxygen saturation will be taken after 5 minutes.

DETAILED DESCRIPTION:
World Health Organization, when systolic blood pressure is equal to or above 130 mm Hg and/or a diastolic blood pressure equal to or above 85 mm Hg , the blood pressure is considered to be raised or high is called hypertension." Most people with hypertension have no symptoms at all; this is why it is known as the "silent killer".

More than 1 in 5 adults worldwide had raised blood pressure. There has been studies on strength exercise, severe aerobic exercise and other types of exercises and on their effects on blood pressure, heart rate and oxygen saturation in other patient populations and on healthy individuals as well, but in the patients with hypertension no comparison has been made between mild and moderate aerobic exercise (tread mill) yet, stating which one is effective. Secondly, already present studies have shown long term effects mostly, not the comparative effects of mild and moderate exercises on blood pressure heart rate and oxygen saturation of patients with hypertension. These techniques are inexpensive, easy to perform and contain no known harmful effect. Hence, current study will undertake this task of finding out what are the comparative effects of mild and moderate aerobic on the BP, heart rate and oxygen saturation and secondly which technique is more effective. Study design will Randomized clinical trial with non-probability convenient sampling.

It will be single blinded study with blinding of assessor. Sample size was calculated from Epitools website and will be 28. There will be two groups which will be randomly assigned 14 people using lottery method. Data will be collected from community dwelling areas of Lahore Patients with hypertension with Systolic Blood Pressure 130 - 159 mmHg and Diastolic Blood Pressure 85 - 99 mmHg (pre hypertensive and stage 1), 30 to 50 years of age, patients who have taken any antihypertensive medicine in more than 6 hours and both males and females will be recruited. Tools will be aneroid sphygmomanometer for measuring blood pressure and pulse oximeter for measuring oxygen saturation and heart rate and Post interventional BP, heart rate readings and oxygen saturation will be taken for both groups on the same day.

Post intervention blood pressure, Heart rate and oxygen saturation will be taken after 5 minutes. Key words: HTN hypertension, HR heart rate, BP blood pressure, vo2max maximum oxygen uptake in unit of time.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 to 55
* Gender: male and female
* Chronic hypertensive stable patients (130 - 159mmHg / 85 - 99mmHg) (3)
* History of hypertension from last 1 year(14)
* Taking anti-hypertensive medicines (ACE inhibitors, calcium channel blockers, thiazide diuretics, ACE receptor inhibitors, beta blockers) more than 6 hours ago

Exclusion Criteria:

History of ischemia

* History of stroke
* Chronic obstructive and restrictive disease
* Hypo and hypernatremia
* Joint disease patients
* Lower limb fracture
* Chronic atrial fibrillation
* Change in drug therapy

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — both male and female are included
Enrollment: 28 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
blood pressure | 6 weeks
  measuring blood pressure by Manual Sphygmomanometer BP apparatus: is the instrument which is used to measure blood pressure if systolic blood pressure is greater than 120 mmHg and diastolic is higher than 90 mmHg is considered hypertensive. Cuff is apply on dominant hand inflate the cuff if sound is appear that is systolic if sound is not hear that is diastolic blood pressure in mmHg.

SECONDARY OUTCOMES:
oxygen saturation | 6 weeks
  measuring oxygen saturation by Pulse oximetry: is the instrument which measure the oxygen saturation and heart rate. Blood Oxygen Saturation (SpO2): The measurement that indicates what percentage of blood is saturated. Normal pulse oximeter readings usually range from 95 to 100 percent. While anything less than 95% indicates underlying medical conditions that need to be evaluated immediately. Pulse Rate / heart rate: Pulse rate is nothing but the heart rate that indicates the number of times a heart beats per minute I.e. 72b/m.
heart rate | 6 weeks
  measuring heart rate by Pulse oximetry: is the instrument which measure the oxygen saturation and heart rate. Blood Oxygen Saturation (SpO2): The measurement that indicates what percentage of blood is saturated. Normal pulse oximeter readings usually range from 95 to 100 percent. While anything less than 95% indicates underlying medical conditions that need to be evaluated immediately. Pulse Rate / heart rate: Pulse rate is nothing but the heart rate that indicates the number of times a heart beats per minute I.e. 72b/m.

CONTACTS AND LOCATIONS:
Overall Officials: Tasneem Shehzadi, Mphil, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clausen JP, Klausen K, Rasmussen B, Trap-Jensen J. Central and peripheral circulatory changes after training of the arms or legs. Am J Physiol. 1973 Sep;225(3):675-82. doi: 10.1152/ajplegacy.1973.225.3.675. No abstract available. PMID 4726503
- [Background] Cao L, Li X, Yan P, Wang X, Li M, Li R, Shi X, Liu X, Yang K. The effectiveness of aerobic exercise for hypertensive population: A systematic review and meta-analysis. J Clin Hypertens (Greenwich). 2019 Jul;21(7):868-876. doi: 10.1111/jch.13583. Epub 2019 Jun 6. PMID 31169988
- [Background] Nascimento LS, Santos AC, Lucena J, Silva L, Almeida A, Brasileiro-Santos MS. Acute and chronic effects of aerobic exercise on blood pressure in resistant hypertension: study protocol for a randomized controlled trial. Trials. 2017 Jun 2;18(1):250. doi: 10.1186/s13063-017-1985-5. PMID 28578691
- [Background] Wen H, Wang L. Reducing effect of aerobic exercise on blood pressure of essential hypertensive patients: A meta-analysis. Medicine (Baltimore). 2017 Mar;96(11):e6150. doi: 10.1097/MD.0000000000006150. PMID 28296729
- [Background] Dimeo F, Pagonas N, Seibert F, Arndt R, Zidek W, Westhoff TH. Aerobic exercise reduces blood pressure in resistant hypertension. Hypertension. 2012 Sep;60(3):653-8. doi: 10.1161/HYPERTENSIONAHA.112.197780. Epub 2012 Jul 16. PMID 22802220
- [Background] Weinstein AA, Chin LM, Keyser RE, Kennedy M, Nathan SD, Woolstenhulme JG, Connors G, Chan L. Effect of aerobic exercise training on fatigue and physical activity in patients with pulmonary arterial hypertension. Respir Med. 2013 May;107(5):778-84. doi: 10.1016/j.rmed.2013.02.006. Epub 2013 Mar 7. PMID 23478192
- [Background] Roque FR, Briones AM, Garcia-Redondo AB, Galan M, Martinez-Revelles S, Avendano MS, Cachofeiro V, Fernandes T, Vassallo DV, Oliveira EM, Salaices M. Aerobic exercise reduces oxidative stress and improves vascular changes of small mesenteric and coronary arteries in hypertension. Br J Pharmacol. 2013 Feb;168(3):686-703. doi: 10.1111/j.1476-5381.2012.02224.x. PMID 22994554
- [Background] Westhoff TH, Schmidt S, Gross V, Joppke M, Zidek W, van der Giet M, Dimeo F. The cardiovascular effects of upper-limb aerobic exercise in hypertensive patients. J Hypertens. 2008 Jul;26(7):1336-42. doi: 10.1097/HJH.0b013e3282ffac13. PMID 18551008
- [Background] Ciolac EG, Guimaraes GV, D'Avila VM, Bortolotto LA, Doria EL, Bocchi EA. Acute aerobic exercise reduces 24-h ambulatory blood pressure levels in long-term-treated hypertensive patients. Clinics (Sao Paulo). 2008 Dec;63(6):753-8. doi: 10.1590/s1807-59322008000600008. PMID 19060996